CLINICAL TRIAL: NCT06111963
Title: Role of Inflammatory Markers Measured Using Flow Cytometry in the Diagnosis and Prognosis of Sepsis in Surgical Cancer Patients
Brief Title: Role of Inflammatory Markers in Sepsis
Status: Completed | Type: Observational
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Assistant Professor of Anesthesia and Pain management, National Cancer Institute, Egypt
Other Study IDs: AP2305-301-001
Record Dates: First submitted 2023-10-16; First posted 2023-11-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Diagnostic
MeSH Terms: conditions — Disease | interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic patients
  Interventions: Diagnostic Test: Serology tests
- Non Septic patients
  Interventions: Diagnostic Test: Serology tests

INTERVENTIONS:
Diagnostic Test: Serology tests — CD4, CD25, IL17

SUMMARY:
A diagnostic and prognostic study, in which the expression of CD64 in activated neutrophils and CD64 and IL17A regulatory T cells in patients with sepsis will be evaluated as a probable marker for sepsis as a primary objective

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients admitted to the surgical ICU following cancer related surgeries and diagnosed with sepsis

Exclusion Criteria:

* Refusal of patient or patient guardian to participate.
* Intraoperative massive blood loss and massive blood transfusion
* Patients with impaired preoperative kidney or liver function tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
To evaluate the expression CD4 | 7 days
  Serology
To evaluate the expression CD25 | 7 days
  Serology
To evaluate the expression IL17 | 7 days
  Serology

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — National Cancer Institute, Cairo University
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt